CLINICAL TRIAL: NCT00971217
Title: Exploring the Effectiveness of the 'Back of the Net' Intervention on Indices of Physical and Psychological Measures
Acronym: BTN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dublin City University (Other)
Responsible Party: Nadine McGale, Dublin City University
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: REC/2009/096
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2011-08-01 (Estimated); Status verified 2011-07

CONDITIONS: Self Concept; Body Fat Composition; Depression; Perceived Social Support
Keywords: Internet based Cognitive-Behavioural Intervention; Exercise Intervention; Depression; Perceived Social Support; Physical Self-Concept
MeSH Terms: conditions — Depression | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Exercise (Experimental): Participants will engage in 2 exercise sessions each week for 10 weeks. Each session will last 50 minutes and will commence with a 5 minute warm up on the bike or treadmill and conclude with a 5 minute cool down. The participants will be required to exercise on their own without interference from others. Participants will wear heart rate monitors to ensure that they are exercising to moderate intensity (70-80% of age predicted maximum heart rate).
  Exercise: Aerobic exercise on the bike/cross trainer/ rower/ treadmill and resistance exercise on the weights machines.
  Interventions: Other: Exercise
- Online Cognitive Behavioural Therapy (Experimental): Participants will be asked to log-on to a web-site specifically aimed at young men once per week and complete the set cognitive-behavioural tasks.
  Interventions: Behavioral: Online Cognitive Behavioural Therapy
- Combined Exercise/Online CBT (Experimental): Participants will simultaneously par-take in both the exercise and the online CBT conditions already outlined.
  Interventions: Other: Exercise; Behavioral: Online Cognitive Behavioural Therapy
- Control (No Intervention): Individuals will be advised that the start of their intervention will be delayed by 10 weeks. After 10 weeks individuals in the control condition will be given the opportunity to avail of an induction session in the gym and subsequently use the gym facilities for three sessions if they so desire. Participants will be asked to refrain from exercise for the 10 week study period.

INTERVENTIONS:
Other: Exercise — Moderate intensity aerobic exercise on the bike/cross trainer/ rower/ treadmill and resistance exercise on the weights machines, twice per week for 10 weeks.
  Other Names: Aerobic exercise
  Arms: Combined Exercise/Online CBT; Exercise
Behavioral: Online Cognitive Behavioural Therapy — Participants will be asked to log-on to a website aimed at young men once per week. Participants will be asked to read a vignette or watch a specific video clip, which will be updated each week by the researcher. Participants will be asked to respond to the vignette/video clip on the website. This should take no longer than 10-15 minutes to complete. Different themes (such as those addressed by traditional cognitive behavioural therapy) will be introduced each week. Themes include: relaxation, identifying positive strengths, body image, goal-setting, problem-solving, resilience, self-care behaviour and sources of support.
  Other Names: 'Back of the Net' Intervention
  Arms: Combined Exercise/Online CBT; Online Cognitive Behavioural Therapy

SUMMARY:
To date very little research has focused on the mental health of young men. The main aim of the proposed research is to explore the effectiveness of a combined exercise and internet-based cognitive behavioral therapy (CBT) intervention (called "Back of the Net") on indices of suicide risk in young men. A second aim is to explore the relationship between physical self-concept, self esteem, body fat composition, body circumference and changes in depression as a result of an exercise intervention. It is hypothesised that the combined exercise and internet-delivered CBT intervention will have greater benefits for indices of suicide risk compared to an exercise-only intervention, an internet-delivered CBT-only intervention and a control condition.

DETAILED DESCRIPTION:
The increase in the number of young people, particularly males, taking their own lives in Ireland has become a major cause for concern. Five times more men than women end their own lives in Ireland today. Research shows that young people, particularly men under 30 years are far less likely to attend their GP than adults aged over 30 years. Thus, young men who are suffering from depression and who are vulnerable to suicidal behaviour are not actively seeking the help they require. Young men are the group least likely to approach mental health services (Russell, Gaffney, Bergin & Bedford, 2004), despite suicide and depression being so prevalent among young Irish males. It is clear that approaches to suicide prevention in Irish society need to bridge the gap between young at-risk men and mental health services.

Research has shown that both psychotherapeutic interventions such as Cognitive Behavioural Therapy (CBT) and exercise interventions can be equally effective as pharmacotherapy in addressing some of the risk factors associated with suicide (Mead et al., 2008), including symptoms of depression. Cognitive-Behavioural Therapy (CBT) places emphasis on identifying and changing maladaptive beliefs and behaviours that contribute to emotional distress. CBT techniques aim to enhance self-control, rational problem-solving abilities and social skills; it is therefore unsurprising that CBT has proven to be beneficial in addressing indices of suicide risk such as depression and perceived social isolation (Barbe, Bridge, Birhamer, Kolko & Brent, 2004; Brown at al., 2005). In an attempt to make CBT more widely available and easily accessible to various populations, research groups are investigating the impact of internet delivered CBT programmes on indices of suicide risk, including depression. Internet delivered CBT programmes have been found to be as effective as face-to-face treatment (Anderson, 2009). Internet delivered CBT has been shown to significantly reduce levels of depression in young people living in Sweden (Anderson, Bergstrom, Hollandare et al., 2005). Research proposes that internet-based interventions represent a paradigm shift in treatment techniques and that internet delivered CBT should be pursued further as a treatment alternative for symptoms of depression (Anderson, 2009; Anderson et al., 2005).

There is a large body of research that supports the role of exercise in treating depressive symptoms. Both depression and feelings of hopelessness, principal indices of suicide, are found to be lower in adults who regularly engage in exercise compared to those who remain sedentary (Chioqueta & Stiles, 2007). In a study involving university students, Chioqueta and Stiles (2007) demonstrate that active engagement in physical activity was significantly associated with improvements in indices of suicide. Involvement in physical activity has been shown to produce positive mood states and subjective well-being as well as reducing stress levels (Fox, 1999).

Suicide prevention in Ireland requires an innovative approach, one that provides support and is easily accessible by young men and which promotes help-seeking behaviour and mental health awareness. It is possible that internet based CBT interventions present such an opportunity for delivering mental health promotion and encouraging help-seeking behaviour among young Irish men while reducing indices of suicide risk. Exercise interventions are similarly successful in reducing the risk factors associated with suicide in young men, such as severity of depressive symptoms. Thus the main aim of this study is to explore the effectiveness of a combined exercise and internet delivered CBT intervention in reducing indices of suicide in young men.

In addition, it has been suggested that Physical Self-Concept mediates the relationship between exercise and self-esteem which is in turn related to depression (Dishman, Hales, Ward et al., 2006). However the relationship between these variables over time as a result of an intervention has not yet been studied. Therefore a secondary aim of this present study is to explore the relationship between physical self-concept, self-esteem and depression throughout the duration of the proposed intervention. We will also examine if changes in body-fat composition and body circumference mediate the relationship between these variables.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged 18-40 years
* Available twice a week for 10 weeks and willing to participate in moderate intensity exercise for 50 minutes at each session
* Not regularly physically active (i.e., engages in a structured exercise session once or less per week)
* Willing to participate in the internet-based CBT intervention once per week for 10 weeks

Exclusion Criteria:

* Current illness or history of clinical conditions that prevents participation in exercise
* Currently alcohol/drug abusing
* Major cognitive or psychiatric impairments
* Currently receiving medication for major psychiatric disorders, including depression

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Depression (Beck Depression Inventory-II). | week 1
Depression (Becks Depression Inventory-II) | week 5
Depression (Becks Depression Inventory-II) | week 10
Depression (Becks Depression Inventory-II) | 8 week follow-up

SECONDARY OUTCOMES:
Perceived Social Support (Social provisions scale) | week 1
Physical Self-Description Questionnaire | week 1
Body Fat Composition | week 1
Body Circumference | week 1
Perceived Social Support (Social provisions scale) | week 5
Perceived Social Support (Social provisions scale) | week 10
Perceived Social Support (Social provisions scale) | 8 week follow-up
Physical Self-Description Questionnaire | week 5
Physical Self-Description Questionnaire | week 10
Physical Self-Description Questionnaire | 8 week follow up
Body Fat Composition | week 5
Body Fat Composition | week 10
Body Fat Composition | 8 week follow up
Body Circumference | week 5
Body Circumference | week 10
Body Circumference | 8 week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nadine McGale, MSc, Principal Investigator — Dublin City University
Locations (1):
- Dublin City University, Dublin, Dublin, Ireland

REFERENCES:
- [Background] Andersson G. Using the Internet to provide cognitive behaviour therapy. Behav Res Ther. 2009 Mar;47(3):175-80. doi: 10.1016/j.brat.2009.01.010. Epub 2009 Feb 20. PMID 19230862
- [Background] Andersson G, Bergstrom J, Hollandare F, Carlbring P, Kaldo V, Ekselius L. Internet-based self-help for depression: randomised controlled trial. Br J Psychiatry. 2005 Nov;187:456-61. doi: 10.1192/bjp.187.5.456. PMID 16260822
- [Background] Barbe RP, Bridge J, Birmaher B, Kolko D, Brent DA. Suicidality and its relationship to treatment outcome in depressed adolescents. Suicide Life Threat Behav. 2004 Spring;34(1):44-55. doi: 10.1521/suli.34.1.44.27768. PMID 15106887
- [Background] Brown GK, Ten Have T, Henriques GR, Xie SX, Hollander JE, Beck AT. Cognitive therapy for the prevention of suicide attempts: a randomized controlled trial. JAMA. 2005 Aug 3;294(5):563-70. doi: 10.1001/jama.294.5.563. PMID 16077050
- [Background] Chioqueta AP, Stiles TC. Cognitive factors, engagement in sport, and suicide risk. Arch Suicide Res. 2007;11(4):375-90. doi: 10.1080/13811110600897143. PMID 17882625
- [Background] Dishman RK, Hales DP, Pfeiffer KA, Felton GA, Saunders R, Ward DS, Dowda M, Pate RR. Physical self-concept and self-esteem mediate cross-sectional relations of physical activity and sport participation with depression symptoms among adolescent girls. Health Psychol. 2006 May;25(3):396-407. doi: 10.1037/0278-6133.25.3.396. PMID 16719612
- [Background] Mead GE, Morley W, Campbell P, Greig CA, McMurdo M, Lawlor DA. Exercise for depression. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD004366. doi: 10.1002/14651858.CD004366.pub3. PMID 18843656
- [Background] Russell V, Gaffney P, Collins K, Bergin A, Bedford D. Problems experienced by young men and attitudes to help-seeking in a rural Irish community. Ir J Psychol Med. 2004 Mar;21(1):6-10. doi: 10.1017/S0790966700008065. PMID 30308724
- [Background] Fox KR. The influence of physical activity on mental well-being. Public Health Nutr. 1999 Sep;2(3A):411-8. doi: 10.1017/s1368980099000567. PMID 10610081